CLINICAL TRIAL: NCT05142774
Title: An Open-Label, Long-Term Extension Study to Evaluate the Safety and Efficacy of Tapinarof Cream, 1% in Subjects With Atopic Dermatitis
Brief Title: Long Term Extension Study of Tapinarof Cream, 1% for Subjects With Atopic Dermatitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DMVT-505-3103
Record Dates: First submitted 2021-10-29; First posted 2021-12-03 (Actual); Results first posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-05

CONDITIONS: Atopic Dermatitis
Keywords: eczema; pediatric; tapinarof; phase 3; topical
MeSH Terms: conditions — Dermatitis, Atopic; Eczema

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- tapinarof cream (Experimental): Subjects entering with vIGA-AD (Validated Investigator Global Assessment of Atopic Dermatitis) ≥1 receive treatment with study drug until they achieve vIGA-AD=0, at which time treatment is discontinued and subjects are monitored for durability of response (remittive response). If/when disease worsening occurs (vIGA-AD ≥2), treatment is re-initiated and continued until vIGA-AD =0 is achieved.
  Subjects entering with a vIGA-AD=0 discontinue treatment and are monitored for duration of remittive response. If/when disease worsening occurs (vIGA-AD ≥2), treatment is re-initiated and continued until vIGA-AD =0 is achieved.
  This treatment and re-treatment pattern of use continue until the end of the study.
  Interventions: Drug: Tapinarof cream, 1%

INTERVENTIONS:
Drug: Tapinarof cream, 1% — Tapinarof cream, 1%, applied daily to affected areas by subjects or their caregivers based on vIGA-AD. Subjects are advised to choose the application time they prefer and apply the study drug at that approximate time each day of study participation.

SUMMARY:
This is an open-label, long-term multicenter, study to evaluate the safety and efficacy of topical tapinarof cream, 1% in subjects with atopic dermatitis. Subjects in this study have completed treatment in one of two Phase 3 pivotal studies (DMVT-505-3101 or DMVT-505-3102) or completed treatment in the DMVT-505-2104 study, or directly enrolled into this study. This study will consist of up to 48 weeks of treatment and a 1 week safety follow-up period.

DETAILED DESCRIPTION:
At the completion of the Week 8 visit of study DMVT-505-3101 (NCT05014568) or study DMVT-505-3102 (NCT05032859) or the Day 28 visit of study DMVT-505-2104 (NCT05186805) (Day 1 [Baseline] in this study), all eligible subjects will be offered enrollment in this open-label long-term extension (OL-LTE) study. Approximately 125 additional pediatric subjects ages 2 to < 18 years who are not eligible for participation in the Phase 3 pivotal studies (DMVT-505-3101 or DMVT-505-3102) will be enrolled directly into this OL-LTE study. Study visits during the treatment period for all subjects will occur every 4 weeks (± 3 days). The total duration of study participation will be approximately 48 weeks for rollover subjects (Baseline to Final Visit) with a 1-week Safety Follow-up Period and approximately 52 weeks for direct-enrolling subjects (Screening to Final Visit) with a 1-week Safety Follow-up Period.

ELIGIBILITY:
Inclusion Criteria:

For Roll-over Subjects Only:

* Met the criteria as a Study Completer in one of three studies (DMVT-505-3101 study, DMVT-505-3102 study, or DMVT-505-2104 study).
* Must not be pregnant at Baseline

For Direct-Enrolling Subjects Only:

* Male and female subjects ages 2 years to < 18 years at the time of consent with clinical diagnosis of AD
* Subjects with a vIGA-AD™ score of ≥ 3 and AD covering ≥ 40% of the BSA at Screening and Baseline (pre-randomization), or subjects with a vIGA-AD™ score of 2 at Screening and Baseline (pre-randomization) regardless of BSA. Subjects must have screened for the DMVT-505-3101 or DMVT-505-3102 study and failed to meet BSA and/or vIGA-AD™ eligibility criteria.
* AD present for at least 6 months for ages 6 years old and above or 3 months for ages 2 to 5 years old
* Must not be pregnant at Screening or Baseline

For All Subjects:

* Female subjects of childbearing potential who are engaging in sexual activity that could lead to pregnancy should use acceptable birth control methods
* Subject, subject's parent, or legal representative must be capable of giving written informed consent/assent

Exclusion Criteria:

For Rollover Subjects Only:

1. Subjects who were not receiving study drug at the time of the last visit in the pivotal study (DMVT-505-3101, DMVT-505-3102, or DMVT-505-2104)
2. Used a prohibited concomitant product or procedure to treat AD during the pivotal study.
3. Had an SAE that was related to treatment or experienced an AE that led to permanent discontinuation of treatment in the pivotal study.
4. Pregnant females

For Direct-Enrolling Subjects:

* Immunocompromised at screening
* Chronic or acute systemic or superficial infection requiring treatment with systemic antibacterials or antifungals within one week prior to baseline visit
* Significant dermatological or inflammatory condition other than AD that, in the Investigator's opinion, would make it difficult to interpret data or assessments during the study
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥2.0x the upper limit of normal (ULN).
* Screening total bilirubin > 1.5x ULN
* Current or chronic history of liver disease
* Current or history of cancer within 5 years except for adequately treated cutaneous basal cell carcinoma, squamous cell carcinoma or carcinoma in situ of the cervix
* Subjects who would not be considered suitable for topical therapy
* Use of any prohibited medication or procedure within the indicated period before the baseline visit including other investigational product within 30 days or 5 half-lives of the investigational product (whichever is longer)
* History of or ongoing serious illness or medical, physical, or psychiatric condition(s) that, in the Investigator's opinion, may interfere with the subject's participation in the study, interpretation of results, or ability to understand and give informed consent.
* Pregnant or lactating females
* History of sensitivity to the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the Investigator or Medical Monitor, contraindicates their participation
* Previous known participation in a clinical study with tapinarof (previously known as GSK2894512 and WBI-1001)

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 728 (Actual)
Dates: Start 2021-10-28 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-03-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Diana Villalobos, Study Director — Dermavant Sciences, Inc.
Locations (101):
- United States (91):
  - Dermavant Investigative Site, Birmingham, Alabama
  - Dermavant Investigative Site, Phoenix, Arizona
  - Dermavant Investigative Site, Scottsdale, Arizona
  - Dermavant Investigative Site, Bryant, Arkansas
  - Dermavant Investigative Site, Fort Smith, Arkansas
  - Dermavant Investigative Site, Cerritos, California
  - Dermavant Investigative Site, Fountain Valley, California
  - Dermavant Investigative Site, Fremont, California
  - Dermavant Investigative Site, Huntington Beach, California
  - Dermavant Investigative Site, Inglewood, California
  - Dermavant Investigative Site, Lancaster, California
  - Dermavant Investigative Site, Long Beach, California
  - Dermavant Investigative Site, Los Angeles, California
  - Dermavant Investigative Site, Mission Viejo, California
  - Dermavant Investigative Site, Sacramento, California
  - Dermavant Investigative Site, San Diego, California
  - Dermavant Investigative Site, San Francisco, California
  - Dermavant Investigative Site, Santa Ana, California
  - Dermavant Investigative Site, Santa Monica, California
  - Dermavant Investigative Site, Thousand Oaks, California
  - Dermavant Investigative Site, Thornton, Colorado
  - Dermavant Investigative Site, Washington D.C., District of Columbia
  - Dermavant Investigative Site, Boca Raton, Florida
  - Dermavant Investigative Site, Brandon, Florida
  - Dermavant Investigative Site, Coral Gables, Florida
  - Dermavant Investigative Site, Delray Beach, Florida
  - Dermavant Investigative Site, Hialeah, Florida
  - Dermavant Investigative Site, Jacksonville, Florida
  - Dermavant Investigative Site, Margate, Florida
  - Dermavant Investigative Site, Miami, Florida
  - Dermavant Investigative Site, Miami Lakes, Florida
  - Dermavant Investigative Site, Orlando, Florida
  - Dermavant Investigative Site, Pinellas Park, Florida
  - Dermavant Investigative Site, Sweetwater, Florida
  - Dermavant Investigative Site, Tampa, Florida
  - Dermavant Investigative Site, Marietta, Georgia
  - Dermavant Investigative Site, Sandy Springs, Georgia
  - Dermavant Investigative Site, Savannah, Georgia
  - Dermavant Investigative Site, Snellville, Georgia
  - Dermavant Investigative Site, Chicago, Illinois
  - Dermavant Investigative Site, Evansville, Indiana
  - Dermavant Investigative Site, Plainfield, Indiana
  - Dermavant Investigative Site, Overland Park, Kansas
  - Dermavant Investigative Site, Lexington, Kentucky
  - Dermavant Investigative Site, Louisville, Kentucky
  - Dermavant Investigative Site, Owensboro, Kentucky
  - Dermavant Investigative Site, Baton Rouge, Louisiana
  - Dermavant Investigative Site, Covington, Louisiana
  - Dermavant Investigative Site, Monroe, Louisiana
  - Dermavant Investigative Site, New Orleans, Louisiana
  - Dermavant Investigative Site, Largo, Maryland
  - Dermavant Investigative Site, Rockville, Maryland
  - Dermavant Investigative Site, Bay City, Michigan
  - Dermavant Investigative Site, Clarkston, Michigan
  - Dermavant Investigative Site, Warren, Michigan
  - Dermavant Investigative Site, Ypsilanti, Michigan
  - Dermavant Investigative Site, New Brighton, Minnesota
  - Dermavant Investigative Site, Missoula, Montana
  - Dermavant Investigative Site, Omaha, Nebraska
  - Dermavant Investigative Site, East Windsor, New Jersey
  - Dermavant Investigative Site, Garden City, New York
  - Dermavant Investigative Site, New York, New York
  - Dermavant Investigative Site, Charlotte, North Carolina
  - Dermavant Investigative Site, Bexley, Ohio
  - Dermavant Investigative Site, Cleveland, Ohio
  - Dermavant Investigative Site, Dayton, Ohio
  - Dermavant Investigative Site, Mason, Ohio
  - Dermavant Investigative Site, Mayfield Heights, Ohio
  - Dermavant Investigative Site, Norman, Oklahoma
  - Dermavant Investigative Site, Oklahoma City, Oklahoma
  - Dermavant Investigative Site, Tulsa, Oklahoma
  - Dermavant Investigative Site, Medford, Oregon
  - Dermavant Investigative Site, Portland, Oregon
  - Dermavant Investigative Site, Anderson, South Carolina
  - Dermavant lnvestigative Site, Greenville, South Carolina
  - Dermavant Investigative Site, Mt. Pleasant, South Carolina
  - Dermavant Investigative Site, North Charleston, South Carolina
  - Dermavant Investigative Site, Spartanburg, South Carolina
  - Dermavant Investigative Site, Knoxville, Tennessee
  - Dermavant Investigative Site, Memphis, Tennessee
  - Dermavant Investigative Site, Bellaire, Texas
  - Dermavant Investigative Site, Cypress, Texas
  - Dermavant Investigative Site, Dallas, Texas
  - Dermavant Investigative Site, Dripping Springs, Texas
  - Dermavant Investigative Site, Grapevine, Texas
  - Dermavant Investigative Site, Houston, Texas
  - Dermavant Investigative Site, San Antonio, Texas
  - Dermavant Investigative Site, Sugar Land, Texas
  - Dermavant Investigative Site, Webster, Texas
  - Dermavant Investigative Site, Richmond, Virginia
  - Dermavant Investigative Site, Spokane, Washington
- Canada (10):
  - Dermavant Investigative Site, Calgary, Alberta
  - Dermavant Investigative Site, Surrey, British Columbia
  - Dermavant Investigative Site, Winnipeg, Manitoba
  - Dermavant Investigative Site, Barrie, Ontario
  - Dermavant Investigative Site, Cobourg, Ontario
  - Dermavant Investigative Site, Oakville, Ontario
  - Dermavant Investigative Site, Ottawa, Ontario
  - Dermavant Investigative Site, Waterloo, Ontario
  - Dermavant Investigative Site, Windsor, Ontario
  - Dermavant Investigative Site, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gold LS, Bruno MJ, Lewitt GM, Hebert AA. Characteristics and management of follicular events and contact dermatitis in patients using tapinarof cream for the treatment of atopic dermatitis or plaque psoriasis. J Dermatolog Treat. 2025 Dec;36(1):2517388. doi: 10.1080/09546634.2025.2517388. Epub 2025 Jul 2. PMID 40600584

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Eligible study participants from DMVT-505-3101 (NCT05014568), DMVT-505-3102 (NCT05032859), and DMVT-505-2104 (NCT05186805) were offered the option of participating in the DMVT-505-3103 open label extension study.
Groups:
- Tapinarof Cream: Tapinarof cream, 1%: Tapinarof cream, 1%, applied daily to affected areas by subjects or their caregivers based on vIGA-AD. Subjects were advised to choose the application time they prefer and apply the study drug at that approximate time each day of study participation.
  Subjects entering with vIGA-AD (Validated Investigator Global Assessment of Atopic Dermatitis) ≥1 received treatment with study drug until they achieved vIGA-AD=0, at which time treatment was discontinued and subjects were monitored for durability of response (remittive response). If/when disease worsening occurs (vIGA-AD ≥2), treatment was re-initiated and continued until vIGA-AD =0 was achieved.
  Subjects entering with a vIGA-AD=0 discontinued treatment and were monitored for duration of remittive response. If/when disease worsening occured (vIGA-AD ≥2), treatment was re-initiated and continued until vIGA-AD =0 was achieved.
  This treatment and re-treatment pattern of use continued until the end of the study.
Period: Overall Study
Arm/Group | Tapinarof Cream
Started | 728
Completed | 497
Not Completed | 231

BASELINE CHARACTERISTICS:
Population: ITT Population
Groups:
- Tapinarof Cream: Subjects entering with vIGA-AD (Validated Investigator Global Assessment of Atopic Dermatitis) ≥1 receive treatment with study drug until they achieve vIGA-AD=0, at which time treatment is discontinued and subjects are monitored for durability of response (remittive response). If/when disease worsening occurs (vIGA-AD ≥2), treatment is re-initiated and continued until vIGA-AD =0 is achieved.
  Subjects entering with a vIGA-AD=0 discontinue treatment and are monitored for duration of remittive response. If/when disease worsening occurs (vIGA-AD ≥2), treatment is re-initiated and continued until vIGA-AD =0 is achieved.
  This treatment and re-treatment pattern of use continue until the end of the study.
  Tapinarof cream, 1%: Tapinarof cream, 1%, applied daily to affected areas by subjects or their caregivers based on vIGA-AD. Subjects are advised to choose the application time they prefer and apply the study drug at that approximate time each day of study participation.
Arm/Group | Tapinarof Cream
Number analyzed (Participants) | 728
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.0 (15.32)
Age, Customized [Count of Participants; unit: Participants]
  2-6 years | 194
  7-11 years | 197
  12-17 years | 213
  ≥18 years | 124
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 389
  Male | 339
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 163
  Not Hispanic or Latino | 562
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4
  Asian | 81
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 219
  White | 383
  More than one race | 27
  Unknown or Not Reported | 13
Region of Enrollment [Number; unit: Count of participants]
  Canada | 112
  United States | 616
Validated Investigator Global Assessment for Atopic Dermatitis [Count of Participants; unit: Participants]
  0 - clear | 58
  1 - almost clear | 189
  2 - mild | 268
  3 - moderate | 182
  4 - severe | 31
Percent Body Surface Area (BSA) [Mean (Standard Deviation); unit: Affected Body Surface Area percentage] | 10.62 (14.259)
Eczema Area and Severity Index (EASI) [Mean (Standard Deviation); unit: units on a scale] | 6.31 (8.247)

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Treatment-Emergent Adverse Events (TEAE) and Serious Adverse Events
Description: For rollover subjects, all AEs reported in this extension study were considered as TEAEs except for those AEs ongoing at the end of previous studies but resolved prior to the Visit 1 date for this extension study. For direct-enrolling subjects, all AEs that start after the first dose of study drug will be considered a TEAE.
Time Frame: Baseline to Week 49
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Tapinarof Cream
Number analyzed (Participants) | 728
Participants
  Any treatment-emergent AE | 451
  Serious treatment-emergent AE | 34

2. Primary Outcome: Frequency of Adverse Events and Serious Adverse Events
Description: All AEs reported in this extension study were considered as TEAEs except for those AEs ongoing at the end of previous studies but resolved prior to the Visit 1 date for this extension study. Subjects could have reported more than one TEAE.
Time Frame: Baseline to Week 49
Population: ITT Population
Measure: Number; unit: Events
Arm/Group | Tapinarof Cream
Number analyzed (Participants) | 728
Events
  Treatment-emergent AE | 1226
  Serious treatment-emergent AE | 45

3. Primary Outcome: Change From Baseline in Clinical Laboratory Values (g/L)
Description: The mean chemistry and hematology parameters were assessed for changes and trends over the course of the study.
Time Frame: Baseline to Week 48
Population: ITT Population, Observed Cases
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Tapinarof Cream
Number analyzed (Participants) | 728
g/L
  Albumin (g/L) | -0.5 (2.43)
  Protein (g/L) | 0.0 (3.95)
  Hemoglobin (g/L) | 1.7 (8.45)
  Ery. Mean Corpuscular HGB Concentration (g/L) | 0.0 (7.61)

4. Primary Outcome: Change From Baseline in Clinical Laboratory Values (U/L)
Description: The mean chemistry parameters were assessed for changes and trends over the course of the study.
Time Frame: Baseline to Week 48
Population: ITT Population, Observed Cases
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Tapinarof Cream
Number analyzed (Participants) | 728
U/L
  Alkaline Phosphatase (U/L) | -14.9 (69.45)
  Alanine Aminotransferase (U/L) | -1.5 (11.96)
  Aspartate Aminotransferase (U/L) | -2.6 (16.13)

5. Primary Outcome: Change From Baseline in Clinical Laboratory Values (mmol/L)
Description: The mean chemistry parameters were assessed for changes and trends over the course of the study.
Time Frame: Baseline to Week 48
Population: ITT Population, Observed Cases
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Tapinarof Cream
Number analyzed (Participants) | 728
mmol/L
  Bicarbonate (mmol/L) | -0.2 (2.31)
  Blood Urea Nitrogen (mmol/L) | 0.04 (1.428)
  Calcium (mmol/L) | -0.019 (0.0926)
  Chloride (mmol/L) | -0.3 (2.43)
  Glucose (mmol/L) | 0.13 (1.462)
  Potassium (mmol/L) | -0.03 (0.493)
  Sodium (mmol/L) | -0.1 (2.14)

6. Primary Outcome: Change From Baseline in Clinical Laboratory Values (Umol/L)
Description: The mean chemistry parameters were assessed for changes and trends over the course of the study.
Time Frame: Baseline to Week 48
Population: ITT Population, Observed Cases
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Tapinarof Cream
Number analyzed (Participants) | 728
umol/L
  Bilirubin (umol/L) | 0.40 (3.434)
  Enzymatic Creatinine (umol/L) | 2.1 (7.92)
  Creatinine (Jaffe) (umol/L) | 2.7 (12.06)
  Urate (umol/L) | 0.9 (52.32)

7. Primary Outcome: Change From Baseline in Clinical Laboratory Values (10^9 Cells/L)
Description: The mean hematology parameters were assessed for changes and trends over the course of the study.
Time Frame: Baseline to Week 48
Population: ITT Population, Observed Cases
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Tapinarof Cream
Number analyzed (Participants) | 728
10^9 cells/L
  Basophils (10^9/L) | 0.01 (0.051)
  Eosinophils (10^9/L) | -.03 (0.308)
  Lymphocytes (10^9/L) | -0.02 (0.909)
  Monocytes (10^9/L) | 0.00 (0.192)
  Neutrophils (10^9/L) | 0.22 (2.079)
  Platelets (10^9/L) | -4.0 (59.57)
  Leukocytes (10^9/L) | 0.18 (2.474)

8. Primary Outcome: Change From Baseline in Clinical Laboratory Values (%)
Description: The mean hematology parameters were assessed for changes and trends over the course of the study.
Time Frame: Baseline to Week 48
Population: ITT Population, Observed Cases
Measure: Mean (Standard Deviation); unit: % of cells
Arm/Group | Tapinarof Cream
Number analyzed (Participants) | 728
% of cells
  Basophils/Total Cells (%) | 0.03 (0.272)
  Eosinophils/Total Cells (%) | -0.39 (3.427)
  Lymphocytes/Total Cells (%) | -0.73 (10.440)
  Monocytes/Total Cells (%) | -0.09 (2.592)
  Neutrophils/Total Cells (%) | 1.18 (11.436)
  Reticulocytes/Erythrocytes (%) | -0.06 (0.402)

9. Primary Outcome: Change From Baseline in Clinical Laboratory Values (L/L)
Description: The hematology parameter, Hematocrit, was assessed for changes and trends over the course of the study.
Time Frame: Baseline to Week 48
Population: ITT Population, Observed Cases
Measure: Mean (Standard Deviation); unit: L/L
Arm/Group | Tapinarof Cream
Number analyzed (Participants) | 728
L/L | 0.005 (0.0263)

10. Primary Outcome: Change From Baseline in Clinical Laboratory Values (pg)
Description: The hematology parameter, Ery. Mean Corpuscular Hemoglobin was assessed for changes and trends over the course of the study.
Time Frame: Baseline to Week 48
Population: ITT Population, Observed Cases
Measure: Mean (Standard Deviation); unit: pg
Arm/Group | Tapinarof Cream
Number analyzed (Participants) | 728
pg | 0.13 (0.823)

11. Primary Outcome: Change From Baseline in Clinical Laboratory Values (fl)
Description: The hematology parameter, Ery. Mean Corpuscular Volume, was assessed for changes and trends over the course of the study.
Time Frame: Baseline to Week 48
Population: ITT Population, Observed Cases
Measure: Mean (Standard Deviation); unit: fl
Arm/Group | Tapinarof Cream
Number analyzed (Participants) | 728
fl | 0.37 (2.364)

12. Primary Outcome: Change From Baseline in Clinical Laboratory Values (10^12 Cells/L)
Description: The hematology parameter, Erythrocytes, was assessed for changes and trends over the course of the study.
Time Frame: Baseline to Week 48
Population: ITT Population, Observed Cases
Measure: Mean (Standard Deviation); unit: 10^12 cells/L
Arm/Group | Tapinarof Cream
Number analyzed (Participants) | 728
10^12 cells/L | 0.038 (0.2905)

13. Primary Outcome: Complete Disease Clearance During LTE: Number of Subjects Achieving Disease Clearance vIGA-AD =0 (Clear) While on Therapy for Subjects Entered LTE vIGA-AD ≥ 1 (Almost Clear )
Description: The vIGA-AD is a clinical tool for assessing the current state/severity of a subject's atopic dermatitis at a given timepoint. It is a static 5-point (0-4) morphological assessment of overall disease severity (scalp excluded), as determined by the investigator, using the clinical characteristics of erythema, induration/papulation, lichenification, oozing/crusting. Higher vIGA-AD scores represents more severe disease.
Time Frame: Baseline to Week 48
Population: ITT Population, Subjects Entering the Study with vIGA-AD Score ≥1, Observed Cases
Measure: Count of Participants; unit: Participants
Arm/Group | Tapinarof Cream
Number analyzed (Participants) | 670
Participants | 320

14. Primary Outcome: Response During LTE: Number of Subjects Achieving vIGA-AD =0 or 1 (Clear or Almost Clear) While on Therapy for Subjects Who Entered LTE With vIGA-AD ≥ 2 (Mild)
Description: as for outcome 13
Time Frame: Baseline to Week 48
Population: ITT Population, Subjects Entering the Study with vIGA-AD Score ≥2, Observed Cases
Measure: Count of Participants; unit: Participants
Arm/Group | Tapinarof Cream
Number analyzed (Participants) | 481
Participants | 347

15. Primary Outcome: Absolute Change From Baseline in %BSA Affected
Description: Subjects received treatment with tapinarof intermittently guided by disease severity. This outcome measure assesses the change from baseline in %BSA affected in all subjects, including those on and those off therapy.
  Assessment of BSA with Atopic Dermatitis was estimated by means of the handprint method, where the full palmar hand of the participant (fully extended palm, fingers and thumb together) represented approximately 1% of the total BSA. Body regions are assigned specific number of handprints with percentage [Head and neck = 10% (10 handprints), upper extremities = 20% (20 handprints), Trunk (including axillae and groin) = 30% (30 handprints), lower extremities (including buttocks) = 40% (40 handprints)]. Lesions on the scalp will not be included in the calculation of %BSA affected. Estimates of the % involvement in each body region will be multiplied by the fraction of total body area to obtain the total %BSA involved by region and overall.
Time Frame: Baseline to Week 48
Population: ITT Population, Observed Cases
Measure: Mean (Standard Deviation); unit: percentage of BSA
Arm/Group | Tapinarof Cream
Number analyzed (Participants) | 506
percentage of BSA | -7.14 (12.881)

16. Primary Outcome: Percent Change From Baseline in %BSA Affected
Description: Subjects received treatment with tapinarof intermittently guided by disease severity. This outcome measure assesses the % change from baseline in %BSA affected in all subjects, including those on and those off therapy.
  Assessment of BSA with Atopic Dermatitis was estimated by means of the handprint method, where the full palmar hand of the participant (fully extended palm, fingers and thumb together) represented approximately 1% of the total BSA. Body regions are assigned specific number of handprints with percentage [Head and neck = 10% (10 handprints), upper extremities = 20% (20 handprints), Trunk (including axillae and groin) = 30% (30 handprints), lower extremities (including buttocks) = 40% (40 handprints)]. Lesions on the scalp will not be included in the calculation of %BSA affected. Estimates of the % involvement in each body region will be multiplied by the fraction of total body area to obtain the total %BSA involved by region and overall.
Time Frame: Baseline to Week 48
Population: ITT Population, Observed Cases; Participants with %BSA=0 at baseline were excluded
Measure: Mean (Standard Deviation); unit: percent change from baseline in % total
Arm/Group | Tapinarof Cream
Number analyzed (Participants) | 462
percent change from baseline in % total | -37.45 (189.905)

17. Primary Outcome: Mean Change From Baseline in Eczema Area and Severity Index (EASI) Score
Description: Subjects received treatment with tapinarof intermittently guided by disease severity. This outcome measure assesses the change from baseline in EASI score in all subjects, including those on and those off therapy.
  The EASI scoring system is a clinical tool that quantifies the severity of a subject's AD based on both lesion severity and %BSA affected. The EASI is a composite score ranging from 0 to 72 that takes into account the degree of erythema, edema/papulation, excoriation, and lichenification (each scored from 0 to 3 separately) for each of four body regions, with adjustment for the %BSA involved for each body region relative to the whole body. The subject's scalp is excluded from this assessment. Higher EASI scores indicate more severe disease.
Time Frame: Baseline to Week 48
Population: ITT Population, Observed Cases
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tapinarof Cream
Number analyzed (Participants) | 506
Units on a scale | -4.19 (7.248)

18. Primary Outcome: Percent Change From Baseline in Eczema Area and Severity Index (EASI) Score
Description: Subjects received treatment with tapinarof intermittently guided by disease severity. This outcome measure assesses the % change from baseline in EASI score in all subjects, including those on and those off therapy.
  The EASI scoring system is a clinical tool that quantifies the severity of a subject's AD based on both lesion severity and %BSA affected. The EASI is a composite score ranging from 0 to 72 that takes into account the degree of erythema, edema/papulation, excoriation, and lichenification (each scored from 0 to 3 separately) for each of four body regions, with adjustment for the %BSA involved for each body region relative to the whole body. The subject's scalp is excluded from this assessment. Higher EASI scores indicate more severe disease.
Time Frame: Baseline to Week 48
Population: ITT Population, Observed Cases; Participants with EASI=0 at baseline were excluded
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tapinarof Cream
Number analyzed (Participants) | 462
Units on a scale | -33.70 (139.557)

19. Primary Outcome: Percent of Subjects With ≥ 50% Improvement in Eczema Area and Severity Index (EASI) From Baseline at Week 48.
Description: The EASI scoring system is a clinical tool that quantifies the severity of a subject's AD based on both lesion severity and %BSA affected. The EASI is a composite score ranging from 0 to 72 that takes into account the degree of erythema, edema/papulation, excoriation, and lichenification (each scored from 0 to 3 separately) for each of four body regions, with adjustment for the %BSA involved for each body region relative to the whole body. Higher EASI scores indicate more severe disease.
Time Frame: Baseline to Week 48
Population: ITT Population, Observed Cases; Participants with EASI=0 at baseline were excluded
Measure: Count of Participants; unit: Participants
Arm/Group | Tapinarof Cream
Number analyzed (Participants) | 462
Participants | 325

20. Primary Outcome: Percent of Subjects With ≥ 75% Improvement in Eczema Area and Severity Index (EASI) From Baseline at Week 48.
Description: The EASI scoring system is a clinical tool that quantifies the severity of a subject's AD based on both lesion severity and %BSA affected. The EASI is a composite score ranging from 0 to 72 that takes into account the degree of erythema, edema/papulation, excoriation, and lichenification (each scored from 0 to 3 separately) for each of four body regions, with adjustment for the %BSA involved for each body region relative to the whole body. The subject's scalp is excluded from this assessment. Higher EASI scores indicate more severe disease.
Time Frame: Baseline to Week 48
Population: ITT Population, Observed Cases; Participants with EASI=0 at baseline were excluded
Measure: Count of Participants; unit: Participants
Arm/Group | Tapinarof Cream
Number analyzed (Participants) | 462
Participants | 256

21. Primary Outcome: Percent of Subjects With ≥ 90% Improvement in Eczema Area and Severity Index (EASI) From Baseline at Week 48.
Description: as for outcome 20
Time Frame: Baseline to Week 48
Population: ITT Population, Observed Cases; Participants with EASI=0 at baseline were excluded
Measure: Count of Participants; unit: Participants
Arm/Group | Tapinarof Cream
Number analyzed (Participants) | 462
Participants | 178

22. Primary Outcome: Mean Change in Peak Pruritis-Numeric Rating Scale (PP-NRS) From Baseline
Description: The Peak Pruritus Numeric Rating Scale (PP-NRS) is used to quickly assess itch/pruritus severity over a 24-hour period. The PP-NRS is scored on a scale of 0 to 10, with 0 being "no itch" and 10 being "worst itch imaginable". The subject or caregiver will utilize the scale to assess peak pruritis once per day and record the results in their diaries. The daily ratings are averaged to generate a score for the week.
Time Frame: Baseline to Week 48
Population: ITT Population, Observed Cases
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tapinarof Cream
Number analyzed (Participants) | 483
Units on a scale | -1.618 (2.7756)

23. Primary Outcome: Number of Subjects With a Baseline Peak Pruritis-Numeric Rating Scale (PP-NRS) Score ≥ 4 Who Achieve ≥ 4-point Reduction in the PP-NRS From Baseline
Description: as for outcome 22
Time Frame: Baseline to Week 48
Population: ITT Population, Subjects with a Baseline PP-NRS Score ≥4, Observed Cases
Measure: Count of Participants; unit: Participants
Arm/Group | Tapinarof Cream
Number analyzed (Participants) | 182
Participants | 94

24. Primary Outcome: Change From Baseline in Vital Signs - Pulse
Description: The mean vital sign parameters were assessed for changes and trends over the course of the study. Shifts from Baseline in vital sign parameters were assessed for clinical relevance.
Time Frame: Baseline to Week 48
Population: ITT Population, Observed Cases
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Arm/Group | Tapinarof Cream
Number analyzed (Participants) | 728
beats per minute (bpm) | -0.9 (12.61)

25. Primary Outcome: Change From Baseline in Vital Signs - Blood Pressure (Systolic and Diastolic)
Description: as for outcome 24
Time Frame: Baseline to Week 48
Population: ITT Population, Observed Cases
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Tapinarof Cream
Number analyzed (Participants) | 728
mmHg
  Systolic Blood Pressure (mmHg) | 1.0 (10.72)
  Diastolic Blood Pressure (mmHg) | 0.7 (9.78)

26. Primary Outcome: Change From Baseline in Vital Signs - Temperature
Description: as for outcome 24
Time Frame: Baseline to Week 48
Population: ITT Population, Observed Cases
Measure: Mean (Standard Deviation); unit: degrees C
Arm/Group | Tapinarof Cream
Number analyzed (Participants) | 728
degrees C | 0.02 (0.437)

ADVERSE EVENTS:
Time Frame: For rollover subjects, all AEs reported in this extension study, through study completion, up to 48 weeks, were considered as TEAEs except for those AEs ongoing at the end of previous studies but resolved prior to the Visit 1 date for this extension study. For direct-enrolling subjects, all AEs that start after the first dose of study drug and through study completion, up to 48 weeks, will be considered a TEAE.
Groups:
- Continuous or Intermittent Use of Tapinarof Cream (DMVT-505) Cream According to vIGA-AD Score: Subjects entering with vIGA-AD (Validated Investigator Global Assessment of Atopic Dermatitis) ≥1 receive treatment with study drug until they achieve vIGA-AD=0, at which time treatment is discontinued and subjects are monitored for durability of response (remittive response). If/when disease worsening occurs (vIGA-AD ≥2), treatment is re-initiated and continued until vIGA-AD =0 is achieved.
  Subjects entering with a vIGA-AD=0 discontinue treatment and are monitored for duration of remittive response. If/when disease worsening occurs (vIGA-AD ≥2), treatment is re-initiated and continued until vIGA-AD =0 is achieved.
  This treatment and re-treatment pattern of use continue until the end of the study.
  Tapinarof cream, 1%: Tapinarof cream, 1%, applied daily to affected areas by subjects or their caregivers based on vIGA-AD. Subjects are advised to choose the application time they prefer and apply the study drug at that approximate time each day of study participation.
Arm/Group | Continuous or Intermittent Use of Tapinarof Cream (DMVT-505) Cream According to vIGA-AD Score
All-Cause Mortality (participants affected / at risk) | 0/728
Serious Adverse Events (participants affected / at risk) | 34/728
Other Adverse Events (participants affected / at risk) | 451/728
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Continuous or Intermittent Use of Tapinarof Cream (DMVT-505) Cream According to vIGA-AD Score (N=728)
Hypothyroidism (Endocrine disorders) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 2 (2)
Pneumonia (Infections and infestations) | 5 (6)
Appendicitis (Infections and infestations) | 1 (1)
Pneumonia respiratory syncytial viral (Infections and infestations) | 1 (1)
Postoperative abscess (Infections and infestations) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Alcohol withdrawal syndome (Psychiatric disorders) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 19 (20)
Status asthmaticus (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dermatitis exfoliative generalised (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Continuous or Intermittent Use of Tapinarof Cream (DMVT-505) Cream According to vIGA-AD Score (N=728)
Vomiting (Gastrointestinal disorders) | 17 (21)
Pyrexia (General disorders) | 16 (19)
Seasonal allergy (Immune system disorders) | 17 (17)
Folliculitis (Infections and infestations) | 88 (101)
Nasopharyngitis (Infections and infestations) | 50 (64)
Upper respiratory tract infection (Infections and infestations) | 50 (73)
COVID-19 (Infections and infestations) | 42 (43)
Influenza (Infections and infestations) | 27 (28)
Impetigo (Infections and infestations) | 22 (26)
Pharyngitis streptococcal (Infections and infestations) | 21 (23)
Ear infection (Infections and infestations) | 17 (24)
Gastroenteritis viral (Infections and infestations) | 17 (18)
Otitis media (Infections and infestations) | 16 (19)
Headache (Nervous system disorders) | 25 (28)
Asthma (Respiratory, thoracic and mediastinal disorders) | 44 (59)
Cough (Respiratory, thoracic and mediastinal disorders) | 24 (27)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-06-16): https://cdn.clinicaltrials.gov/large-docs/74/NCT05142774/Prot_000.pdf
  • Statistical Analysis Plan (2023-04-21): https://cdn.clinicaltrials.gov/large-docs/74/NCT05142774/SAP_001.pdf